CLINICAL TRIAL: NCT03807791
Title: Study of Prevalence and Risk Factors of Hypovitaminosis C in Long Term Care Unit
Acronym: Vitamin C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL18_0392
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Vitamin C Deficiency; Scurvy
Keywords: Vitamine C deficiency; skin rash; scurvy; food texture; geriatric institution; Unit Of Long Term Care
MeSH Terms: conditions — Ascorbic Acid Deficiency; Scurvy; Exanthema | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient living in the Unit of Long Term Care (Experimental): Patient living in the Unit of Long Term Care without any limit time
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — A blood sample will be taken by the nurse of our unit within a week after their consent. It consists as a simple blood sample and it will be taken during the normal analysis planed by the chief of the service in order to avoid to collect two different samples.
  The measurement method will use equipment from the Lyon Sud hospital laboratory. The samples need a pre-treatment in the 3 hours after taking the blood to avoid the oxidation of vitamin C and a result lower than expected.

SUMMARY:
The clinical finding of skin rashes which appear after a vitamin C deficiency in Long Term Care Unit leads us to believe that the institutional diet could predispose to this kind of deficiency. Vitamin C has a key role into the struggle against oxidant stress and is involved into the connective tissue formation of the skin and the vascular endothelium. Vitamin C deficiency affects currently 15 to 25% of the elderly over 65 years old reaching 15% women and 20% men after 65 according to Johnston and Al. It concerns mainly the people in precarious situations (persons without fixed homes, ethyl-smoking persons) and elderly over 65 years. Hypovitaminosis C, defined by plasma level between 5 mg/L and 15 mg/L (28.41 to 85.23 µmol/L), is currently undiagnosed, especially with people with a risk of food deficiency and its prevalence increases with age. The treatment consists of a daily oral supplementation of 1 gram of vitamin C/d for 15 days. A minimum intake of 10 mg/D of vitamin C is required to prevent scurvy and maintain a total pool of 350 mg. A diet modification by a systematic intake of 2 glasses of fresh orange juice and/or the consumption of raw fruits and vegetables would prevent the appearance of scurvy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 65 years old
* living in the Unit of Long Term Care without any limit time.
* with a system of social insurance
* Who gave its consent by his own , or with help of his representant or his tutor or curator.

Exclusion Criteria:

* rejection of the blood sample
* patient feeding with articial nutritional feeding (stomach tube feeding)
* person close to death, who is not able to feed himself and / or with life-threatening in short time.
* Patient with personal history of vitamin C deficiency.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Vitamin C plasma level | Between day 0 and day 7.
  1. ) Collection of the consent
  2. ) At the same time as other analysis for current cares a blood sample taken by a nurse of our unit to determine plasma levels of vitamin C.
  3. ) Registration of risk factors of vitamin C deficiency. .
  4. ) Doing a clinical exam within 7 days after the blood sample.

SECONDARY OUTCOMES:
Supposed risk factors of hypovitaminosis C | Day 0
  The supposed risk factors are represent by general risk factors, Anthropometric parameters, Nutritional risk factors, Risk factors because of Unit of Long Term Care, Pathologies associated, Clinical signs associated with vitamin C deficiency
Cutaneous symptoms | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de soins Longue Durée, Hôpital Pierre Garraud (Hospices Civils de Lyon), Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lagorsse C., Oumédian E., Bourguignon L, de La Gastine B. Les carences en vitamine C, une cause peu connue d'affections cutanées en institution gériatrique : à propos de 2 cas en Unité de Soins de Longue Durée (USLD). Rev Geriatr 2019 Février 44 2.